CLINICAL TRIAL: NCT00621192
Title: Multiple Dose Pharmacokinetic Study of Meropenem in Young Infants (<91 Days) With Suspected or Complicated Intra-abdominal Infections
Brief Title: Pharmacokinetic (PK) and Safety Study of Meropenem in Young Infants With Intra-abdominal Infections
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: The Emmes Company, LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HHSN267200700051C; HHSN267200700051C (Other: NICHD)
Record Dates: First submitted 2008-02-20; First posted 2008-02-22 (Estimated); Results first posted 2011-11-29 (Estimated); Last update posted 2023-04-25 (Actual); Status verified 2023-03

CONDITIONS: Necrotizing Enterocolitis; Intra-abdominal Infection
Keywords: meropenem; infants; intra-abdominal infection; pharmacokinetics; safety
MeSH Terms: conditions — Enterocolitis, Necrotizing; Intraabdominal Infections | interventions — Meropenem

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Meropenem (Experimental): These
  Participants were subdivided into the following four groups based on Gestational Age (GA) and Postnatal Age (PNA):
  Group 1: GA at birth below 32 weeks - PNA <2 weeks; Group 2: GA at birth below 32 weeks - PNA ≥2 weeks and <91 days; Group 3: GA at birth 32 weeks or older - PNA <2 weeks; Group 4: GA at birth 32 weeks or older - PNA ≥2 weeks and <91 days.
  Interventions: Drug: meropenem

INTERVENTIONS:
Drug: meropenem — Meropenem was administered concomitantly with compatible medications. Because an in-line filter is not appropriate due to drug binding, the 30 minute infusion was rate controlled by using appropriate infusion (syringe) pumps. Dosing and administration of other antimicrobial therapy (e.g., an aminoglycoside) was administered per local standard of care at the discretion of the infant's neonatologist. If there was a delay in the study drug shipment, sites were to use open-label meropenem to protect the safety of the participant.
  20 mg/kg every 12 hours in infants <32 weeks GA and PNA < 2 weeks 20 mg/kg every 8 hours in infants <32 weeks GA and PNA ≥ 2 weeks 20 mg/kg every 8 hours in infants ≥32 weeks GA and PNA < 2 weeks 30 mg/kg every 8 hours in infants ≥32 weeks GA and PNA ≥ 2 weeks
  Other Names: Merrem

SUMMARY:
Meropenem is an antibiotic that is commonly used to treat serious infections. Although it is used in premature and young infants, the correct dose is not known. The purpose of this study is to determine the correct dose and the safety of meropenem for the treatment of complicated intra-abdominal infections in these young babies.

DETAILED DESCRIPTION:
This study will evaluate the safety, tolerability and Pharmacokinetics - Pharmacodynamics (PK-PD) of meropenem in infants <91 days of age with suspected and complicated intra-abdominal infections.

The specific aims of this trial are:

1. To characterize meropenem single-dose and multiple-dose PK in subjects with suspected and complicated intra-abdominal infections.
2. To characterize the safety profile of meropenem in the treatment of suspected and complicated intra-abdominal infections.
3. To assess collected efficacy data for meropenem for the treatment of suspected and complicated intra-abdominal infections.

ELIGIBILITY:
Inclusion Criteria:

1. Written permission from parent or legal guardian
2. Age younger than 91 days
3. Likely to survive beyond the first 48 hours after enrollment
4. Sufficient intravascular access (either peripheral or central) to receive study drug.

   AND ONE OF THE FOLLOWING
5. 1) Physical, radiological, and/or bacteriological findings of a complicated intra-abdominal infection. These include peritonitis, NEC (Necrotizing Enterocolitis) Grade II or higher by Bell's criteria, Hirschsprung's disease with perforation, spontaneous perforation, meconium ileus with perforation, bowel obstruction with perforation, as evidenced by free peritoneal air on abdominal radiograph, intestinal pneumatosis or portal venous gas on abdominal radiographic examination.

OR 2) Possible NEC OR 3) Otherwise receiving meropenem per local standard of care

Exclusion criteria:

1. Renal dysfunction evidenced by urine output <0.5 mL/hr/kg over the prior 24 hours
2. Serum creatinine >1.7 mg/dL
3. History of clinical seizures or EEG (Electroencephalogram) confirmed seizures
4. Concomitant treatment with another carbapenem (ertapenem or imipenem) at the time of informed consent
5. Any condition which would make the subject or the caregiver, in the opinion of the investigator, unsuitable for the study

Max Age: 90 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 200 (Actual)
Dates: Start 2008-06; Primary Completion 2009-10 (Actual); Study Completion 2009-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Danny Benjamin, MD, PhD, MPH, Principal Investigator — Duke University
Locations (26):
- United States (26):
  - University of Alabama, Birmingham, Alabama
  - Children's Hospital of Oakland, Oakland, California
  - Children's Hospital of Orange County, Orange, California
  - University of California Medical Center, San Diego, California
  - Sharp-Mary Birch Hospital for Women, San Diego, California
  - Yale New Haven Hospital, New Haven, Connecticut
  - Children's National Medical Center, Washington D.C., District of Columbia
  - University of Florida, Gainesville, Florida
  - Kapiolani Medical Center for Women and Children, Honolulu, Hawaii
  - Evanston Northwestern Healthcare, Evanston, Illinois
  - Indiana University - Riley Hospital for Children, Indianapolis, Indiana
  - University of Louisville, Louisville, Kentucky
  - University of Michigan, Ann Arbor, Michigan
  - Kansas City Children's Mercy Hospital, Kansas City, Missouri
  - Albany Medical Center, Albany, New York
  - Suny Downstate Medical Center, Brooklyn, New York
  - Duke University Medical Center, Durham, North Carolina
  - Duke University, Durham, North Carolina
  - Akron Children's Hospital, Akron, Ohio
  - Case Western Reserve, RB&C, UHCMC, Cleveland, Ohio
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Magee Women's Hospital, Pittsburgh, Pennsylvania
  - Vanderbilt Children's Hospital, Nashville, Tennessee
  - University of Texas Southwestern Medical Center, Dallas, Texas
  - Baylor College of Medicine, Houston, Texas
  - University of Utah medical Center, Salt Lake City, Utah

REFERENCES:
- [Derived] Cohen-Wolkowiez M, Poindexter B, Bidegain M, Weitkamp JH, Schelonka RL, Randolph DA, Ward RM, Wade K, Valencia G, Burchfield D, Arrieta A, Mehta V, Walsh M, Kantak A, Rasmussen M, Sullivan JE, Finer N, Rich W, Brozanski BS, van den Anker J, Blumer J, Laughon M, Watt KM, Kearns GL, Capparelli EV, Martz K, Berezny K, Benjamin DK Jr, Smith PB; Meropenem Study Team. Safety and effectiveness of meropenem in infants with suspected or complicated intra-abdominal infections. Clin Infect Dis. 2012 Dec;55(11):1495-502. doi: 10.1093/cid/cis758. Epub 2012 Sep 5. PMID 22955430

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Enrollment Period - June 19, 2008 to October 6, 2009 Locations - Hospitals including University Hospitals Total number of sites - 24 Total number of participants - 200
Pre-assignment Details: Other antimicrobials in addition to meropenem was used in the study due to concerns regarding the safety and ethics of using monotherapy in this patient population.The study was designed as an open-label, dose escalation study because sufficient data regarding the feasibility of a randomized, active controlled efficacy study was unavailable.
Groups:
- 1. GA <32 Wks; PNA<2 Wks: Group 1: GA at birth below 32 weeks - PNA < 2 weeks;
- 2. GA <32 Wks; PNA 91days ≥ 2Wks: Group 2: GA at birth below 32 weeks - PNA ≥ 2 weeks and < 91 days
- 3. GA ≥ 32 Wks; PNA <2 Wks: Group 3: GA at birth 32 weeks or older - PNA < 2 weeks;
- 4. GA ≥32 Wks; PNA 91 Days ≥ 2 Wks: Group 4: GA at birth 32 weeks or older - PNA ≥ 2 weeks and < 91 days.
Period: Overall Study
Arm/Group | 1. GA <32 Wks; PNA<2 Wks | 2. GA <32 Wks; PNA 91days ≥ 2Wks | 3. GA ≥ 32 Wks; PNA <2 Wks | 4. GA ≥32 Wks; PNA 91 Days ≥ 2 Wks
Started | 39 | 103 | 31 | 27
Safety Population | 39 | 103 | 31 | 27
Efficacy Population | 39 | 101 | 28 | 27
Completed | 35 | 94 | 26 | 24
Not Completed | 4 | 9 | 5 | 3
Not completed — Withdrawal by Subject | 0 | 0 | 2 | 0
Not completed — Physician Decision | 1 | 3 | 0 | 0
Not completed — Protocol Violation | 1 | 0 | 0 | 1
Not completed — Adverse Event | 0 | 1 | 0 | 1
Not completed — Death | 2 | 5 | 0 | 0
Not completed — Final Assessments not Completed | 0 | 0 | 3 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | 1. GA <32 Wks; PNA<2 Wks | 2. GA <32 Wks; PNA 91days ≥ 2Wks | 3. GA ≥ 32 Wks; PNA <2 Wks | 4. GA ≥32 Wks; PNA 91 Days ≥ 2 Wks | Total
Number analyzed (Participants) | 39 | 103 | 31 | 27 | 200
Age, Continuous [Mean (Standard Deviation); unit: Days] — Post Natal Age (in days)
  Days
    Mean Postnatal Age | 8.5 (3.3) | 38.3 (19.3) | 6.5 (3.5) | 36.0 (22.0) | 27.3 (21.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15 | 47 | 9 | 11 | 82
  Male | 24 | 56 | 22 | 16 | 118
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 5 | 16 | 4 | 3 | 28
  Not Hispanic or Latino | 32 | 81 | 27 | 24 | 164
  Unknown or Not Reported | 2 | 6 | 0 | 0 | 8
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 1 | 0 | 1 | 2
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 1 | 0 | 2
  Black or African American | 12 | 33 | 8 | 5 | 58
  White | 25 | 65 | 21 | 18 | 129
  More than one race | 1 | 2 | 0 | 2 | 5
  Unknown or Not Reported | 0 | 2 | 1 | 1 | 4

OUTCOME MEASURES:

1. Primary Outcome: Efficacy Success (Alive at Efficacy Visit,Last Culture (if Obtained) From Sterile Body Fluid is Negative for Bacteria (Except Staphylococcus Species) From Start of Study Drug Until Efficacy Visit,Presumptive Clinical Cure Score(PCCS) >7 at Efficacy Visit)
Description: The PCCS was derived by comparing clinical signs and symptoms prior to administration of the first dose of study drug and study Day 28.The elements of the PCCS include Mean BP,Temp,PaO2(mmHg)/FiO2,Lowest serum pH,seizures,Urine output,Cardiovascular inotrope support,C-reactive protein (CRP)and Abdominal girth.
  Score - Asymptomatic to Asymptomatic 1;Asymptomatic to Worsening 0;Symptomatic to Worsening 0;Symptomatic to No change 0;Symptomatic to Improved 1;Symptomatic to Asymptomatic 1
  If 7 or more of 10 signs received a score of 1, then the infant was considered a presumptive clinical cure.
  GA stands for Gestational Age and PNA stands for Postnatal Age.
Time Frame: Average of 12 days (3 to 21 days)
Population: The Efficacy Population includes all patients who have efficacy assessment (Clinical Signs) at Pre-Dose and Study Day 28 (or the day that the Day 28 assessments were taken).
Measure: Number; unit: Participants
Arm/Group | 1. GA <32 Wks; PNA<2 Wks | 2. GA <32 Wks; PNA 91days ≥ 2Wks | 3. GA ≥ 32 Wks; PNA <2 Wks | 4. GA ≥32 Wks; PNA 91 Days ≥ 2 Wks
Number analyzed (Participants) | 39 | 98 | 28 | 27
Participants | 29 | 82 | 26 | 25

2. Primary Outcome: Deaths
Time Frame: Up to 51 days (Recorded from the time of informed consent until 72 hours following the last dose of study drug)
Population: The Safety Population includes all patients who receive any amount of meropenem.
Measure: Number; unit: Participants
Arm/Group | 1. GA <32 Wks; PNA<2 Wks | 2. GA <32 Wks; PNA 91days ≥ 2Wks | 3. GA ≥ 32 Wks; PNA <2 Wks | 4. GA ≥32 Wks; PNA 91 Days ≥ 2 Wks
Number analyzed (Participants) | 39 | 103 | 31 | 27
Participants | 3 | 8 | 0 | 0

3. Primary Outcome: Meropenem Clearance
Description: Given the limited availability of blood for Pharmacokinetic (PK) assessments in this population a sparse sampling approach was utilized. Subjects were assigned to one of two Dose 1 sample collection schedules, "PK-odd" and "PK-even" based on birth date to ensure collection of PK data throughout the dose interval. In addition, PK samples were collected around approximately the 5th dose. Subjects that did not have Dose 1 PK samples could have steady-state (Dose 5) using the Dose 5 PK collection schedule.
Time Frame: Up to 7-8hrs post drug administration
Measure: Mean (Standard Deviation); unit: L/h/kg
Arm/Group | 1. GA <32 Wks; PNA<2 Wks | 2. GA <32 Wks; PNA 91days ≥ 2Wks | 3. GA ≥ 32 Wks; PNA <2 Wks | 4. GA ≥32 Wks; PNA 91 Days ≥ 2 Wks
Number analyzed (Participants) | 39 | 98 | 28 | 27
L/h/kg | 0.089 (0.027) | 0.122 (0.037) | 0.135 (0.040) | 0.202 (0.061)

4. Primary Outcome: Key Safety Endpoints
Description: Safety assessments included death, seizure documentation (including correlation of serum meropenem level and seizures), strictures, perforation, wound dehiscence, short gut, development of extended beta lactamase infection, development of candidiasis, antimicrobial therapy failure
Time Frame: Up to 51 days (Adverse Events (AEs) were recorded from the time of informed consent until 72 hours following the last dose of study drug)
Population: Safety Population - The Safety Population includes all patients who receive any amount of meropenem.
Measure: Number; unit: Participants
Arm/Group | 1. GA <32 Wks; PNA<2 Wks | 2. GA <32 Wks; PNA 91days ≥ 2Wks | 3. GA ≥ 32 Wks; PNA <2 Wks | 4. GA ≥32 Wks; PNA 91 Days ≥ 2 Wks
Number analyzed (Participants) | 39 | 103 | 31 | 27
Participants
  Death | 3 [1.6% to 20.9%] | 8 | 0 | 0
  Seizure | 4 | 3 | 1 | 2
  Strictures | 0 | 0 | 0 | 0
  Perforation | 2 | 2 | 0 | 0
  Wound Dehiscence | 1 | 1 | 1 | 1
  Development of Candidiasis | 5 | 3 | 0 | 0
  Antimicrobial Therapy Failure | 7 | 12 | 2 | 2

ADVERSE EVENTS:
Time Frame: Adverse Events (AEs) were recorded from the time of informed consent until 72 hours following the last dose of study drug for non-Serious Adverse Events (SAEs) and until 30 days after the last dose of study drug for SAEs.
Description: Any AE that occurred between the time informed consent was obtained and the initial dose of study, that was considered related to a protocol specified procedure, were reported.
  The Investigator was responsible for assessing relationship of AE to study medication using the following definitions:Not related, possibly, probably or definitely related.
Arm/Group | 1. GA <32 Wks; PNA<2 Wks | 2. GA <32 Wks; PNA 91days ≥ 2Wks | 3. GA ≥ 32 Wks; PNA <2 Wks | 4. GA ≥32 Wks; PNA 91 Days ≥ 2 Wks
Serious Adverse Events (participants affected / at risk) | 9/39 | 18/103 | 2/31 | 5/27
Other Adverse Events (participants affected / at risk) | 9/39 | 8/103 | 2/31 | 3/27
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 1. GA <32 Wks; PNA<2 Wks (N=39) | 2. GA <32 Wks; PNA 91days ≥ 2Wks (N=103) | 3. GA ≥ 32 Wks; PNA <2 Wks (N=31) | 4. GA ≥32 Wks; PNA 91 Days ≥ 2 Wks (N=27)
Bradycardia (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Congenital diaphragmatic Hernia (Congenital, familial and genetic disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Patent Ductus Arteriosus (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Retinopathy of Prematurity (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Colonic Stenosis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Illeal Perforation (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Intestinal Ischaemia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Intestinal Obstruction (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Intestinal perforation (Gastrointestinal disorders) | 2 (2) | 2 (2) | 0 (0) | 0 (0)
Intestinal Stenosis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Necrotising Colitis (Gastrointestinal disorders) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Rectal Haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Multi-organ failure (General disorders) | 2 (2) | 2 (2) | 0 (0) | 0 (0)
Abdominal Sepsis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Bacterial Sepsis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Fungal Sepsis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Meningitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Respiratory Synctial Virus Infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Sepsis (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Wound Dehiscence (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Chest X-Ray Abnormal (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Subarachnoid Haemorrhage (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Apnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pneumonia Aspiration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pulmonary Haemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Respiratory Arrest (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Respiratory Distress (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 1. GA <32 Wks; PNA<2 Wks (N=39) | 2. GA <32 Wks; PNA 91days ≥ 2Wks (N=103) | 3. GA ≥ 32 Wks; PNA <2 Wks (N=31) | 4. GA ≥32 Wks; PNA 91 Days ≥ 2 Wks (N=27)
Sepsis (Infections and infestations) | 5 (12) | 5 (12) | 1 (12) | 1 (12)
Convulsion (Nervous system disorders) | 4 (10) | 3 (10) | 1 (10) | 2 (10)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No